CLINICAL TRIAL: NCT02803918
Title: Randomized, Double-blind, Placebo-controlled, Dose Escalation, Study on Safety, Pharmacokinetics and Pharmacodynamics of Lixisenatide in Pediatric Patients With Type 2 Diabetes Mellitus Not Adequately Controlled With Metformin and/or Basal Insulin
Brief Title: A Study on Safety, Pharmacokinetics and Pharmacodynamics of Lixisenatide in Pediatric Patients With Type 2 Diabetes Mellitus (T2DM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TDR14311; U1111-1176-6142 (Other: UTN)
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lixisenatide; Metformin

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lixisenatide (Experimental): Administration of 3 ascending repeated doses of lixisenatide once daily and subcutaneously. Background therapy (metformin and basal insulin) will be administered daily about the same time as usually done.
  Interventions: Drug: Lixisenatide (AVE0010); Drug: Basal Insulin; Drug: Metformin
- Placebo (Placebo Comparator): Administration of 3 ascending repeated doses of matching placebo once daily and subcutaneously. Background therapy (metformin and basal insulin) will be administered daily about the same time as usually done.
  Interventions: Drug: Placebo; Drug: Basal Insulin; Drug: Metformin

INTERVENTIONS:
Drug: Lixisenatide (AVE0010) — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Arms: Lixisenatide
Drug: Placebo — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Arms: Placebo
Drug: Basal Insulin — Pharmaceutical form: solution
  Route of administration: subcutaneous
Drug: Metformin — Pharmaceutical form: tablet
  Route of administration: oral

SUMMARY:
Primary Objective:

To demonstrate safety of 14-day repeated lixisenatide doses with 3 ascending doses as compared to placebo in pediatric patients with T2DM.

Secondary Objectives:

* To evaluate plasma concentrations of lixisenatide after repeated doses (3 ascending doses) and pharmacokinetic parameters of repeated lixisenatide doses in pediatric patients with T2DM.
* To evaluate the change from baseline in fasting and post-prandial plasma glucose concentrations during a standardized meal test after 3 ascending repeated doses of lixisenatide in comparison to placebo.

DETAILED DESCRIPTION:
The total study duration will be up to 10 weeks that includes a 6-week treatment period with dose escalation every 2 weeks.

ELIGIBILITY:
Inclusion criteria :

* Male or female patients aged ≥10 and <18 years old (at least 4 patients below 16 years old).
* Body mass index (BMI) >85th percentile for age and gender; BMI ≤50 kg/m2.
* Male and female patients with documented T2DM insufficiently controlled with metformin at a stable dose and regimen for 8 weeks prior to randomization and/or basal insulin at stable dose (± 20%) and regimen for 8 weeks prior to randomization. The exact individual metformin dose will be selected according to local regulation and to the investigator's medical judgment.
* Glycated hemoglobin (HbA1c) >6.5% and ≤11% at screening.

Exclusion criteria:

* If female, ongoing pregnancy (defined as positive serum pregnancy test), breast-feeding.
* Sexually active postmenarchal female patient who does not agree to use an adequate and highly effective method of contraception throughout the study duration and according to local regulation (ie, hormonal contraception, condom, etc.).
* Diabetes other than T2DM.
* Fasting plasma glucose >250 mg/dL (>13.9 mmol/L) at screening.
* Use of other oral or injectable antidiabetic or hypoglycemic agents other than metformin and basal insulin (eg, alpha glucosidase inhibitor, glucagon-like peptide (GLP-1) receptor agonist, dipeptidyl peptidase-IV (DPP-IV) inhibitors, short-acting insulin etc.) within 1 month prior to the screening visit.
* History of unexplained pancreatitis, chronic pancreatitis, pancreatectomy, stomach/gastric surgery, inflammatory bowel disease.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events (AEs) | Up to 10 weeks
Number of patients with treatment-emergent adverse events (TEAEs) | Up to 10 weeks
Number of patients with anti-lixisenatide antibodies | Up to 10 weeks

SECONDARY OUTCOMES:
Assessment of pharmacokinetic (PK) parameters: lixisenatide plasma concentration | Day 14, Day 28 and Day 42
Assessment of PK parameters: maximum concentration (Cmax) | Day 42
Assessment of PK parameters: time to reach Cmax (Tmax) | Day 42
Assessment of PK parameters: area under up to last concentration (AUClast) | Day 42
Assessment of PK parameters: area under curve (AUC) | Day 42
Assessment of pharmacodynamic parameter: plasma glucose AUC-0-4.5 hours | Day 14, Day 28 and Day 42

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (11):
- United States (4):
  - Investigational Site Number 840002, Baton Rouge, Louisiana
  - Investigational Site Number 840006, New Orleans, Louisiana
  - Investigational Site Number 840009, Philadelphia, Pennsylvania
  - Investigational Site Number 840007, Lufkin, Texas
- Investigational Site Number 480001, Phoenix, Mauritius
- Mexico (2):
  - Investigational Site Number 484001, Monterrey
  - Investigational Site Number 484002, Puebla City
- Investigational Site Number 710001, Cape Town, South Africa
- Investigational Site Number 724002, Barcelona, Spain
- Turkey (Türkiye) (2):
  - Investigational Site Number 792002, Ankara
  - Investigational Site Number 792001, Izmir

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Barrientos-Perez M, Hsia DS, Sloan L, Nell H, Mungur O, Hovsepian L, Schmider W, Spranger R, Yang N, Niemoeller E. A study on pharmacokinetics, pharmacodynamics and safety of lixisenatide in children and adolescents with type 2 diabetes. Pediatr Diabetes. 2022 Sep;23(6):641-648. doi: 10.1111/pedi.13343. Epub 2022 Apr 24. PMID 35411611